CLINICAL TRIAL: NCT05850715
Title: Translation, Cross-cultural Adaptation, Reliability and Validity of the Greek Version of the Disability Assessment for Dementia Scale (DAD-Gr)
Brief Title: Cross-cultural Adaptation of the Greek Version of Disability Assessment for Dementia
Acronym: DAD-Gr
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Georgios Marios Kyriakatis, Undergraduate Student, Department of Physiothrapy, School of Health Sciences, University of Thessaly
Other Study IDs: 416, 30/3/2023
Record Dates: First submitted 2023-03-31; First posted 2023-05-09 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Disability Assessment for Dementia (DAD) — The scale consists of 40 items and assesses patients' independence in basic and instrumental activities. The scale is completed by the patient's caregiver with the assistance of the assessor-therapist.

SUMMARY:
The main purpose of this study is primarily the translation and cross-cultural adaptation into Greek and then the investigation of validity and reliability in the Greek target population.

DETAILED DESCRIPTION:
Two investigators will do the translation into Greek, then a third person independent of the first two will translate the scale backward, i.e. into English. Then, the three investigators will meet with another independent investigator who is familiar with the field of Greek translations of foreign language rating scales. Thus, the final translation and Greek version of the scale will be created. Then, the process of finding the participants will begin and the first assessment with the scale will be carried out initially. After two days will take place reassessment for the reliability of the measurement tool. In order to find the validity of the scale in the Greek population, in the first assessment will be used also Katz index for Basic Activities of Daily Living and the Lawton scale for Instrumental Activities of Daily Living.

ELIGIBILITY:
Inclusion Criteria:

* be diagnosed with any type of dementia
* have a carer
* have a good cognitive level

Exclusion Criteria:

* be end-stage or bedridden

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include patients with dementia of good cognitive level and necessarily have a caregiver. Patients may also live independently or with relatives or in a public or private care facility.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Disability Assessment for Dementia and change from baseline | At baseline and after two days for checking the change and therefore the reliability. The score can range between 0 - 40, where 40 means complete independence in activities of daily living.
  The scale is completed by the patient's caregiver with the assistance of the assessor-therapist.

SECONDARY OUTCOMES:
Katz index for Basic Activities of Daily Living | At baseline. The score can range between 0 - 6, where 6 means complete independence in basic activities of daily living.
  The scale consists of 6 questions and will be asked to the caregiver by the assessor.
Lawton scale for Instrumental Activities of Daily Living | At baseline.The score can range between 0 - 8 for women and 0 - 5 for men, where the highest scores means complete independence in basic activities of daily living.
  The scale consists of 8 questions and will be asked to the caregiver by the assessor.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Besios, Dr., Study Director — Assistant Professor
Locations (1):
- University of Thessaly, Lamia, Fthiotis, Greece

REFERENCES:
- [Background] Gelinas I, Gauthier L, McIntyre M, Gauthier S. Development of a functional measure for persons with Alzheimer's disease: the disability assessment for dementia. Am J Occup Ther. 1999 Sep-Oct;53(5):471-81. doi: 10.5014/ajot.53.5.471. PMID 10500855
- [Background] Sanchez-Perez A, Lopez-Roig S, Perez AP, Gomez PP, Pastor MA, Pomares MH. Validation Study of the Spanish Version of the Disability Assessment for Dementia Scale. Medicine (Baltimore). 2015 Nov;94(44):e1925. doi: 10.1097/MD.0000000000001925. PMID 26554794
- [Background] Tozlu M, Cankurtaran M, Yavuz BB, Cankurtaran ES, Kutluer I, Erkek BM, Halil M, Ulger Z, Cosgun E, Ariogul S. Functional disability in Alzheimer disease: a validation study of the Turkish version of the disability assessment for dementia scale. J Geriatr Psychiatry Neurol. 2014 Dec;27(4):237-46. doi: 10.1177/0891988714532014. Epub 2014 Apr 24. PMID 24763071